CLINICAL TRIAL: NCT06386445
Title: Study on the Serum Metabolic Markers and Early Complications After Allogeneic Hematopoietic Stem Cell Transplantation in Hemaotological Diseases： Cohort Study
Brief Title: Study on the Serum Metabolic Markers and Early Complications After Allo-HSCT： Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF-CRF-2023-XK013
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Stem Cell Transplant Complications; Acute Graft Versus Host Disease; Acute Kidney Injury; Major Adverse Cardiac Events
MeSH Terms: conditions — Acute Kidney Injury; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- XJTU Cohort of allo-HSCT: all the patients underwent allogeneic stem cell transplantation
  Interventions: Other: Serum metabolomics sequencing

INTERVENTIONS:
Other: Serum metabolomics sequencing — Serum samples from the day before pre-treatment, day after pre-treatment, 2 weeks，4 weeks，8 weeks and 12 weeks after transplantation will be detected by metabolomics sequencing.

SUMMARY:
This study aims to establish a cohort of 500 patients with hematological disease who undergoing allogeneic hematopoietic stem cell transplantation in the northwest region. All patients will be followed up at the outpatient clinic once a week after transplantation until 100 days after transplantation to observe the presence of acute graft versus host disease, acute kidney damage, and major cardiovascular adverse events. Serum samples from the day before pre-treatment, day after pre-treatment, 2 weeks，4 weeks，8 weeks and 12 weeks after transplantation will be detected by metabolomics sequencing.The primary objective is to explore the serum metabolic markers of acute graft versus host disease，acute kidney injury, and major adverse cardiac events within 100 days after transplantation，the secondary objective is to observe the high-risk factors for early complications.

DETAILED DESCRIPTION:
This study aims to establish a cohort of 500 patients with hematological disease who undergoing allogeneic hematopoietic stem cell transplantation in the northwest region. All patients will be followed up at the outpatient clinic once a week after transplantation until 100 days after transplantation to observe the presence of acute graft versus host disease, acute kidney damage, and major cardiovascular adverse events. Baseline characterisitcs of patients, including gender, age, disease type, transplant type, donor gender and age, pre-transplant baseline electrocardiogram, myocardial enzymology, renal function, and other indicators were recorded. Serum samples from the day before pre-treatment, day after pre-treatment, 2 weeks，4 weeks，8 weeks and 12 weeks after transplantation will be detected by metabolomics sequencing.The primary objective is to explore the serum metabolic markers of acute graft versus host disease，acute kidney injury, and major adverse cardiac events within 100 days after transplantation，the secondary objective is to observe the high-risk factors for early complications.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 65 years old;

Gender unlimited;

Normal heart and kidney function before transplantation;

Patients with indications for allogeneic hematopoietic stem cell transplantation.

Exclusion Criteria:

* CREA or BUN higher than the normal upper limit value before transplantation;

Individuals with a history of arrhythmia, heart failure, or PCI stent implantation prior to transplantation;

Patients with mental illness;

Those who are unwilling to sign informed consent.

Ages: 0 Years to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hematological disease underwent allogeneic stem cell transplantation
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
acute graft versus host disease | within 100 days after transplantation
  skin，liver and gastrointestinal acute graft versus host disease

SECONDARY OUTCOMES:
acute kidney injury | within 100 days after transplantation
  Included AKI-R, AKI-I, and AKI-F ，the criteria for classification of AKI-R, AKI-I, and AKI-F are as follows: AKI-R was considered if there was an increase in serum creatinine to more than 1.5-fold of baseline value or a urinary output lower than 0.5 ml/kg/h for 6 h. AKI-I was considered if there was an increase in serum creatinine to more than 2-fold of baseline value or urinary output lower than 0.5 ml/kg/h for 12 h. AKI-F was considered if there was an increase in serum creatinine to more than 3-fold baseline value or urinary output lower than 0.3 ml/kg/h for 24 h.
major adverse cardiac events | within 100 days after transplantation
  cardiovascular mortality, coronary events, heart failure, atrial fibrillation/flutter

CONTACTS AND LOCATIONS:
Overall Officials: pengcheng he, M.D., Study Director — First Affiliated Hospital Xi'an Jiaotong University

IPD SHARING:
Plan to Share IPD: No